CLINICAL TRIAL: NCT00694187
Title: A Single Dose, Two-Period, Two-Treatment, 2-Way Crossover Bioequivalency Study of Zaleplon 10 mg Capsules Under Fasting Conditions.
Brief Title: Bioequivalency Study of Zaleplon 10 mg Capsules Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, DRA-MA, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZALE-01
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Short Term Treatment of Insomnia
MeSH Terms: interventions — zaleplon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Zaleplon

SUMMARY:
The objective of this study was to show the bioequivalence of a Roxane Laboratories' Zaleplon Capsules, 10 mg, to Sonata ® Capsules, 10 mg (Jones Pharma) under fasting conditions using a single-dose, randomized, 2-treatment, 2-period, 2-sequence crossover design

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to Zaleplon or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2004-01; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Baseline, Two Period, Seven day washout

CONTACTS AND LOCATIONS:
Overall Officials: So Ran Hong, M.D., Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, Houston, Texas, United States